CLINICAL TRIAL: NCT02086266
Title: The Efficacy of Pilates Compared to Pelvic Floor Muscle Training Associated With Electrical Stimulation in the Recovery of Post-prostatectomy Urinary Incontinence: a Randomized Clinical Trial.
Brief Title: The Efficacy of Pilates in the Recovery of Post-prostatectomy Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Fabiana Rotondo Pedriali, Physioterapist student of a masters degree program at the Center of Health Science, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PILUI1
Record Dates: First submitted 2014-03-09; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer; Urinary Incontinence
Keywords: Prostatectomy; Urinary Continence; Physical Therapy Modalities; Pelvic Floor; Randomized Trial.
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — Exercise Movement Techniques

ARMS (2):
- PILATES (Experimental): Weekly Pilates sessions, guided by a specialized physiotherapist. The duration of the treatment was 10 weeks, and each session lasted 45 to 50 minutes. All subjects received instruction to perform specific daily home exercises.
  Interventions: Other: PILATES
- PFMT and AES (Active Comparator): For also 10 weeks, the participants went trough anal electrical stimulation associated with Pelvic Floor Muscle Training, supervised by a specialized physiotherapist. All subjects received orientation to perform the same pelvic floor exercises at home.
  Interventions: Other: PFMT and AES

INTERVENTIONS:
Other: PILATES
  Arms: PILATES
Other: PFMT and AES
  Arms: PFMT and AES

SUMMARY:
The purpose of this study is to compare the efficacy between a Pilates exercise program and a Pelvic Floor Muscle Training (PFMT) protocol combined with anal electrical stimulation (AES) in the recovery of urinary continence (UI) after radical prostatectomy.

There are no studies that evaluate Pilates mat exercises for incontinence in men although it can be assured that this method has the pelvic floor contractions as a principle for practice. If this new therapeutic approach proves to be as effective as described treatment in improving urinary complaints, it will be an option for patients who prefer a non-invasive treatment.

DETAILED DESCRIPTION:
This randomized clinical trial includes 69 individuals with urinary incontinence one month after radical prostatectomy. One physiotherapist, with experience in urogynecology, was responsible for all the assessments. Urinary frequency, nocturia, 24-hour pad test, number of pads used per day, and the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) were the variables evaluated.

The subjects were allocated in one of two treatment groups (G1: Pilates; G2: anal electrical stimulation combined with pelvic floor muscle training). Volunteers participated of 10 sessions of the corresponding treatment and were reassessed objectively by the number of pads used per day, and subjectively with the score of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 50 and 75 years old;
* Submitted to radical prostatectomy;
* With complaints of urinary incontinence;
* That completed one month of surgery;

Exclusion Criteria:

* History of incontinence;
* Transurethral resection of the prostate;
* Diagnosis of neurological or cognitive impairment;
* Subjects who were unable to attend treatment sessions, due to distance or physical limitations.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in the number of pads used per day at 3 months | 3 months

SECONDARY OUTCOMES:
Change in the 24 hours Pad Test at 3 months | 3 months
Change in the International Consultation of Urinary Incontinence- Short Form at 3 months | 3 months
Change in the episodes of nocturia at 3 months | 3 months

REFERENCES:
- [Derived] Johnson EE, Mamoulakis C, Stoniute A, Omar MI, Sinha S. Conservative interventions for managing urinary incontinence after prostate surgery. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD014799. doi: 10.1002/14651858.CD014799.pub2. PMID 37070660